CLINICAL TRIAL: NCT03558191
Title: A Single-arm, Open Label, Multi-center, Phase 2 Study of SHR-1210 in Recurrent/Metastatic Nasopharyngeal Carcinoma Patients Who Have Received Previous At Least Two Lines of Chemotherapy.
Brief Title: SHR-1210 in Recurrent/Metastatic Nasopharyngeal Carcinoma Who Have Received Previous At Least Two Lines of Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-209
Record Dates: First submitted 2018-05-30; First posted 2018-06-15 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Recurrent/Metastatic Nasopharyngeal Carcinoma; PD-1
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 Injection (Experimental): SHR-1210 injection, 200 mg/dose, intravenous infusion over 30 minutes, once every 2 weeks .
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — A humanized monoclonal immunoglobulin PD-1 antibody
  Other Names: Camrelizumab

SUMMARY:
This is an open label, single-arm, multi-center, phase 2 Study of SHR-1210 in recurrent/metastatic nasopharyngeal carcinoma(R/M NPC) patients who have received previous at least two lines of chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this phase 2 study is to assess objective response rate of SHR-1210 in patients with R/M NPC. The secondary objective is to observe the duration of response, progression free survival, time to response, overall survival and safety of SHR-1210 in R/M NPC. ADA is also investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Recurrent/Metastatic Nasopharyngeal Carcinoma (WHO type II-III);
2. Stage IVb R/M NPC failed from first-line platinum based chemotherapy and second-line chemotherapy;
3. ECOG performance status of 0 or 1;
4. Life expectancy ≥ 12 weeks;
5. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria;
6. Can provide either a newly obtained or archival tumor tissue sample;
7. Adequate laboratory parameters during the screening period as evidenced by the following:

   1. Absolute neutrophil count ≥ 1.5 × 10^9/L ;
   2. Platelets ≥ 90 × 10^9/L;
   3. Hemoglobin ≥ 9.0 g/dL;
   4. Serum albumin ≥ 2.8g/dL;
   5. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), ALT and AST ≤ 1.5×ULN
   6. Creatinine clearance≥50 mL/min;
8. Female of child bearing potential, a negative urine or serum pregnancy test result within 72 h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 60 days after the last dose of SHR-1210. Male subjects with WOCBP partner must be willing to use adequate contraception for the course of the study through 120 days after the last dose of SHR-1210;
9. Subjects must be willing to participate in the research and sign an informed consent form (ICF);

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease;
2. Subjects having clinical symptoms of metastases to central nervous system (such as cerebral edema, requiring steroids intervention, or brain metastasis progression);
3. Has a known additional malignancy within the last 5 years before study treatment with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers;
4. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
5. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy;
6. Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy within 4 weeks prior to first dosing or not recovered to ≤CTCAE 1 from adverse events (except for hair loss or neurotoxic sequelae from prior platinum therapy) due to a previously administered agent. Palliative irradiation should be ended 2 weeks before first dosing;
7. Active infection or an unexplained fever > 38.5°C before two weeks of first dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
8. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C;
9. Currently participating or has participated in a study within 4 weeks of the first dose of study medication;
10. Received a live vaccine within 4 weeks of the first dose of study medication. Pregnancy or breast feeding;
11. Received a systematic antibiotics within 4 weeks of the first dose of study medication.

    Pregnancy or breast feeding.
12. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent;
13. Subjects are known to have a history of psychiatric substance abuse, alcoholism, or drug addiction;
14. Pregnancy or breast feeding;
15. According to the investigator, other conditions that may lead to stop the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Cancer Center of Sun-Yat Sen University (CCSYSU); Qing Yang, MD, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao BJ, Sima XX, Chen G, Gulizeba H, Zhou T, Huang Y. Predictive and prognostic role of early apolipoprotein A-I alteration in recurrent or metastatic nasopharyngeal carcinoma patients treated with anti-PD-1 therapy. Cancer Med. 2023 Aug;12(16):16918-16928. doi: 10.1002/cam4.6321. Epub 2023 Jul 6. PMID 37409613

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHR-1210 Injection
Started | 156
Treated | 156
Completed | 131
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 149
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 156
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 156

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assess by Independent Review Committee (IRC)
Description: Percentage of participants achieved partial response (PR) or complete response (CR) based on IRC assessment according to the RECIST (version 1.1) is presented for this endpoint.
  Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks (28 days) after the criteria for response are first met. Only tumor assessments performed on or before the start date of any further anti-cancer therapies are considered in the assessment of best overall response .
Time Frame: Tumor assessments were conducted at every 8 weeks from the first dose until the end of treatment, withdrawal of consent, or death ，whichever was earlier, approximately 3 years.
Population: The primary efficacy endpoint was analyzed in FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
percentage of participants | 28.3 [21.3 to 36.2]

2. Secondary Outcome: ORR Assess by Investigators
Description: Percentage of participants achieved partial response (PR) or complete response (CR) based on investigator assessment according to the RECIST (version 1.1) is presented for this endpoint.
  Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks (28 days) after the criteria for response are first met. Only tumor assessments performed on or before the start date of any further anti-cancer therapies are considered in the assessment of best overall response.
Time Frame: Tumor assessments were conducted at every 8 weeks from the first dose until the end of treatment, withdrawal of consent, or death (whichever was earlier), approximately 3 years.
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
percentage of participants | 24.3 [17.8 to 32.0]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined, for participants with a CR or PR per RECIST version 1.1, as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or death, whichever occurs first.
Time Frame: as for outcome 2
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
month | 20.3 [13.0 to 30.5]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants achieving PR, CR or SD (SD ≥ 8 weeks) based on IRC assessment according to the RECIST version 1.1 is presented in this endpoint. DCR is a best overall response from the time of first dose to the documented objective progression or the subsequent anti-tumor therapy (whichever occurs first).
Time Frame: as for outcome 2
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
percentage of participants | 54.6 [46.3 to 62.7]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the first dose to the date of the first documentation of PD or death, whichever occurs first. PFS was based on investigator assessment according to the RECIST version 1.1. PFS time was summarized using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
month | 3.7 [2.0 to 5.4]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from the first dose to death due to any cause. OS time was measured using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: The secondary efficacy endpoint was analyzed in FAS.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SHR-1210 Injection
Number analyzed (Participants) | 152
month | 18.7 [15.2 to 20.1]

ADVERSE EVENTS:
Time Frame: AEs should be reported from the time the participant has taken at least 1 dose of study treatment through the participant's last visit (approximately 3 years).
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | SHR-1210 Injection
All-Cause Mortality (participants affected / at risk) | 11/156
Serious Adverse Events (participants affected / at risk) | 37/156
Other Adverse Events (participants affected / at risk) | 154/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Injection (N=156)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
pulmonary inflammation (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
progressive disease (General disorders) | 7
fever (General disorders) | 3
infectious pneumonia (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
anemia (Blood and lymphatic system disorders) | 2
Reactive capillary hyperplasia (Immune system disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 1
Chest Discomfort (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Bacterial pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
elevated GGT (Investigations) | 1
elevated blood bilirubin (Investigations) | 1
Increased creatine phosphokinase (Investigations) | 1
elevated blood alkaline phosphatase (Investigations) | 1
decreased platelet count (Investigations) | 1
Brain radiation Injury (Injury, poisoning and procedural complications) | 1
Radiation osteonecrosis (Injury, poisoning and procedural complications) | 1
Infusion-related reactions (Injury, poisoning and procedural complications) | 1
Dysphagia (Gastrointestinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Squamous cell carcinoma of tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Injection (N=156)
Anaemia (Blood and lymphatic system disorders) | 82
Hypothyroidism (Endocrine disorders) | 42
Constipation (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 10
Pyrexia (General disorders) | 39
Asthenia (General disorders) | 35
Chest discomfort (General disorders) | 14
Chest pain (General disorders) | 14
Reactive capillary endothelial proliferation (Immune system disorders) | 140
Upper respiratory tract infection (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 9
Aspartate aminotransferase increased (Investigations) | 47
White blood cell count decreased (Investigations) | 37
Alanine aminotransferase increased (Investigations) | 30
Occult blood positive (Investigations) | 25
Blood thyroid stimulating hormone increased (Investigations) | 22
Gamma-glutamyltransferase increased (Investigations) | 16
Neutrophil count decreased (Investigations) | 15
Blood creatinine increased (Investigations) | 14
Urinary occult blood positive (Investigations) | 14
Thyroxine free decreased (Investigations) | 13
Weight decreased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 11
Platelet count decreased (Investigations) | 11
Blood lactate dehydrogenase increased (Investigations) | 10
Bilirubin conjugated increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 31
Decreased appetite (Metabolism and nutrition disorders) | 25
Hyponatraemia (Metabolism and nutrition disorders) | 21
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 17
Hypoaesthesia (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 13
Proteinuria (Renal and urinary disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 51
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 26
Rash (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03558191/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT03558191/SAP_001.pdf